CLINICAL TRIAL: NCT07139223
Title: The Effect of Laughter Yoga on Premenstrual Syndrome Symptoms and Quality of Life in Young Women: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Premenstrual Syndrome Symptoms and Quality of Life in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Gülsüm Akkuş, Lecturer, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LokmanHekimU-KDH-GA-01
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: Premenstrual Syndrome-PMS
Keywords: Premenstrual Syndrome; Laughter Yoga; Quality of Life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, randomized, parallel-group controlled trial with a 1:1 allocation ratio. Eligible participants will be randomly assigned to either the intervention group (laughter yoga sessions twice a week for 4 weeks, followed by 4 weeks of structured daily individual laughter practices) or the control group (no intervention during the study period). Assessments will be conducted at baseline, after the 4-week group sessions, and after the 8-week follow-up. The primary outcome is the change in PMS symptom severity, and the secondary outcome is the change in quality of life. Due to the nature of the intervention, participants and providers cannot be blinded; however, data will be coded and analyzed by a statistician blinded to group allocation
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and intervention providers cannot be blinded. However, the statistician performing the data analysis will remain blinded to group allocation. Data will be coded, and the statistician will analyze the outcomes without knowledge of whether participants belong to the intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): Intervention arm: Laughter yoga group sessions will be implemented twice a week for 4 weeks (8 sessions in total); the first session will be ~45 min, the subsequent sessions ~30 min. Sessions will be conducted face-to-face in a suitable room within the institution. Following the interim measurement in week 4, the intervention arm will continue structured individual laughter practices daily for 4 weeks.
  Interventions: Behavioral: laughter yoga
- control arm (No Intervention): No intervention will be applied to the control arm; after the post-tests, the same training will be offered to this group for ethical reasons (delayed intervention).

INTERVENTIONS:
Behavioral: laughter yoga — Intervention arm: Laughter yoga group sessions will be implemented twice a week for 4 weeks (8 sessions in total); the first session will be ~45 min, the subsequent sessions ~30 min. Sessions will be conducted face-to-face in a suitable room within the institution. Following the interim measurement in week 4, the intervention arm will continue structured individual laughter practices daily for 4 weeks.
  Arms: intervention arm

SUMMARY:
Premenstrual syndrome (PMS) is a common condition among young women, characterized by physical, emotional, and behavioral symptoms that negatively affect quality of life. Laughter yoga, a non-pharmacological mind-body intervention combining breathing techniques, relaxation, and intentional laughter, has been shown to reduce stress, improve mood, and enhance well-being. This randomized controlled trial aims to evaluate the effect of laughter yoga on PMS symptoms and quality of life in young women.

DETAILED DESCRIPTION:
The menstrual cycle is a physiological process that begins at puberty and continues until menopause. PMS is a recurrent condition that occurs in the luteal phase of the cycle and subsides with menstruation. It is associated with a wide range of psychological, physical, and behavioral symptoms, including irritability, depression, breast tenderness, bloating, sleep disturbances, and decreased academic or social functioning. These symptoms significantly impair daily activities and reduce quality of life, particularly in young women.

The prevalence of PMS varies across populations, but studies consistently indicate that approximately half of young women experience moderate to severe symptoms. In some cases, these symptoms result in absenteeism, reduced productivity, and academic difficulties. The most severe form, premenstrual dysphoric disorder (PMDD), affects a smaller proportion of women but has a profound impact on functioning.

Management of PMS includes both pharmacological and non-pharmacological interventions. Pharmacological treatments such as oral contraceptives, antidepressants, and hormonal therapies may provide relief but often cause side effects and are not always preferred by young women. Non-pharmacological approaches, including relaxation techniques, exercise, yoga, and complementary therapies, are increasingly considered due to their accessibility and fewer side effects.

Laughter yoga is a mind-body practice developed in the 1990s, combining breathing exercises, playful activities, and simulated laughter that soon turns into genuine laughter. The brain does not distinguish between spontaneous and voluntary laughter, and both can induce positive physiological and psychological effects. Research has shown that laughter yoga reduces stress, enhances immune function, increases endorphins, and promotes overall well-being. It is a simple, cost-effective, and sustainable intervention that can be applied individually or in groups.

Although laughter yoga has been studied in relation to stress reduction, mood enhancement, and chronic disease management, there is limited evidence regarding its specific effects on PMS. Preliminary findings suggest potential benefits in reducing PMS-related distress, but no randomized controlled trial has comprehensively examined its impact on both PMS symptoms and quality of life.

This randomized controlled trial is designed to address this gap. The intervention group will participate in structured laughter yoga sessions guided by a certified instructor, while the control group will receive no intervention during the study period. PMS symptom severity and quality of life will be assessed using validated scales at baseline, during the intervention, and at follow-up.

The study aims to provide scientific evidence on the effectiveness of laughter yoga as a non-pharmacological approach in PMS management. By evaluating both short-term and sustained effects, this trial seeks to contribute to women's health literature with an innovative, low-cost, and accessible intervention. The findings are expected to inform clinical practice and support the integration of laughter yoga into nursing and women's health care for improving symptom management and quality of life in young women.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing premenstrual symptoms (PMS score of 110 or higher),
* Are between the ages of 18-25,
* Have regular menstrual periods,
* Can read and understand Turkish,

Exclusion Criteria:

* Students who completed the pretest data collection forms incompletely,
* Students who were taking medication due to a chronic illness,
* Students who were using hormonal contraceptive methods,
* Students who had any health problems that could create a communication barrier,
* Students who were receiving medication for insomnia (such as SSRIs and SNRIs),
* Students who were receiving treatment for PMS,
* Students who were pregnant or lactating in the last 12 months,
* Students who exercised regularly (affecting homogeneity between groups and intervention effectiveness),
* Students who had a diagnosed psychiatric illness (depression, panic attacks, schizophrenia, etc.),
* Students who had a condition that prevented them from practicing laughter yoga (abdominal surgery within the last three months, uncontrolled hypertension, glaucoma, hernia, epilepsy).

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The reason why only female participants were included in the study is that premenstrual syndrome is a syndrome that occurs only in women.
Enrollment: 69 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Symptom Severity | 8 week
  The Premenstrual Syndrome Scale (PMS) will be used to assess participants. Participants will first take a pre-intervention pretest. They will then complete a total of eight laughter yoga sessions twice a week for four weeks. Interim measurements will be taken after the laughter yoga sessions are completed. Participants will be assigned homework assignments to practice laughter practices daily for four weeks. Following the homework assignments, a post-test will be administered to assess changes in PMS symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Didem ŞİMŞEK KÜÇÜKKELEPÇE, Study Director — Lokman Hekim University
Locations (1):
- Bilecik Seyh Edebali University, Bilecik, Bir Eyalet Seçin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No